CLINICAL TRIAL: NCT01773278
Title: Cholesterol and Antioxidant Treatment in Patients With Smith-Lemli-Opitz Syndrome (SLOS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-410
Record Dates: First submitted 2012-12-03; First posted 2013-01-23 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Smith-Lemli-Opitz Syndrome; Cone-Rod Dystrophy; Hearing Loss
Keywords: Antioxidant treatment; Oxysterols; Cholesterol deficiency; Accumulation of 7-dehydrocholesterol; electroretinogram (ERG); Auditory Brainstem Response (ABR)
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome; Cone-Rod Dystrophies; Hearing Loss | interventions — Antioxidants; Cholesterol; Eggs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- antioxidant effects on retinal function (Experimental): Patients with SLOS will be treated with both cholesterol supplementation and antioxidants. Retinal function will be followed by serial electroretinogram (ERG) testing and pigmentary retinopathy will be followed by Serial Ophthalmologic exams under anesthesia
  Interventions: Drug: Antioxidants; Drug: Cholesterol
- antioxidant effects on hearing (Experimental): Patients with SLOS will be treated with cholesterol and antioxidant medication and their hearing will be followed by serial brainstem audiometry (ABR)
  Interventions: Drug: Antioxidants; Drug: Cholesterol
- Antioxidant effect on Oxysterols (Experimental): Patients with SLOS will be treated with antioxidants and cholesterol. Blood oxysterol levels will be measured. Future focus will be on being able to use oxysterol levels to regulate antioxidant doses, and to determine which particular antioxidants might have the most benefit in lowering oxysterols
  Interventions: Drug: Antioxidants; Drug: Cholesterol

INTERVENTIONS:
Drug: Antioxidants — Patients will be prescribed the drug DEKAS plus at a dose based on age and weight. The effects of the treatment will be monitored by serial ERG, ABR, oxysterol levels and clinical findings. Blood levels of 25-Oh vitamin D will be monitored to prevent toxicity.
  Other Names: DEKAS Plus
Drug: Cholesterol — Patients with SLOS typically have cholesterol deficiency. They will be treated with cholesterol supplementation to keep cholesterol levels > 100 mg/dl if possible
  Other Names: cholesterol suspension; eggs; Slo-lesterol

SUMMARY:
Patients with biochemically confirmed SLOS are being treated with cholesterol supplementation and antioxidant medication. They are carefully monitored with visits to clinic, laboratory testing including cholesterol and 7-dehydrocholesterol levels, vitamin levels, blood counts and liver and kidney function. On a serial basis, no more often than once a year, the patients undergo a series of tests under anesthesia, including electroretinogram (ERG), brainstem audiometry (ABR), and ophthalmologic exam under anesthesia to follow pigmentary retinopathy.

DETAILED DESCRIPTION:
Smith-Lemli-Opitz Syndrome (SLOS) is an autosomal recessive disorder caused by a metabolic error in the final step of cholesterol biosynthesis, leading to cholesterol deficiency and accumulation of the cholesterol precursor, 7-dehydrocholesterol.Patients with SLOS display complex medical problems including growth failure, intellectual disability, behavioral disorders, progressive retinal dystrophy, hearing loss and photosensitivity. Dr Elias was one of the original geneticists who discovered the cause of this disorder in 1994, and ever since has been treating SLOS patients with cholesterol supplementation. In 2008, a second medication called AquADEKS, a mixture of vitamins and other compounds with antioxidant properties was added to the treatment regimen. AquADEKS has since been replaced with a comparable medication named DEKAS plus.The purpose of the DEKAS plus is to allow treatment with antioxidant medications in an effort to prevent retinal degeneration, hearing and skin problems associated with SLOS.

This protocol has been approved by the Colorado Multiple Institutional Review Board and supported by the Clinical Translational Research Center (CTRC) since 2001. The following updated information is available about the protocol:

1. Research has revealed that oxysterols are toxic compounds made from the cholesterol precursor, 7-dehydrocholesterol. These oxysterol compounds are severely neurotoxic and toxic to the retina, and treatment with antioxidants may help lower their levels, resulting in slowing of retinal deterioration. Testing of oxysterol levels in patients with SLOS is now ongoing, in collaboration with a laboratory at University of Washington in Seattle (Dr Libin Xu). It is hoped that testing of oxysterol levels in blood may help provide more updated info to help guide treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Smith-Lemli-Opitz Syndrome
* Elevated levels of 7-dehydrocholesterol and 8-dehydrocholesterol
* Must be able to travel to Children's Hospital Colorado annually
* Must have insurance coverage for ERG/ABR studies

Exclusion Criteria:

* absence of detectable 7-dehydrocholesterol/8-dehydrocholesterol
* allergy to Antioxidant medication

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-12; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Electroretinogram (ERG) results over time | 1-2 year
  ERG testing will be performed on an serial basis while the patient is being treated with antioxidants (AquADEKS), to follow the amplitude and latency time on ERG. Improvement would be determined by an increased amplitude and decreased latency time.

SECONDARY OUTCOMES:
Change in ABR (Auditory Brainstem response) testing over time | 1-2 years
  Patients will be followed serial with ABR to determine the latency time in Wave I, when treated with antioxidant medication

OTHER OUTCOMES:
Change in Blood Oxysterol measurements over time | 12-24 months
  Oxysterols can be measured in blood specimens from SLOS patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Elias, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No